CLINICAL TRIAL: NCT00870285
Title: Ustekinumab Plus UVB-311nm Half-side Phototherapy in Patients With Psoriasis
Brief Title: Ustekinumab Plus UVB-311nm in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Graz IRB 20-253 ex 08/09
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biologic; Ustekinumab; UVB-311nm narrowband; phototherapy; half-side comparison
MeSH Terms: conditions — Psoriasis | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: UVB 311nm radiation — UVB-311nm radiation given 3 times a week to one randomized body-half
  Other Names: narrow-band UVB radiation

SUMMARY:
Ustekinumab, an IL-12/23 antibody has been approved in the E.C. and U.S.A. for the treatment of moderate to severe psoriasis. The aim of this study is to determine in a randomized half-side comparison whether additional narrowband UVB-311nm phototherapy accelerates and improves the clearance of skin lesions in Ustekinumab-treated patients.

DETAILED DESCRIPTION:
Patients with moderate to severe psoriasis who receive standard treatment with Ustekinumab (45 mg at week 0, 4, and every 12 weeks) are exposed to UVB-311nm phototherapy on a randomized body half (left or right; head exempt) 3 x per week for six weeks and/or until complete response (defined as reduction in PASI to < 3). PASI score, patient visual analogue score (VAS) for therapeutic response, and patient VAS for severity of skin lesions is assessed weekly; and at follow-up visits at month 3, 6, and 12. Paired Wilcoxon testing for differences in PASI and patient VAS scores is done; Fischer exact test is applied to determine differences in complete remission, PASI reduction > 90%, > 75% and/or 50% between body sites.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Psoriasis patients who receive treatment with Ustekinumab

Exclusion Criteria:

* Age below 18 years
* Pregnancy or lactation
* History of malignant melanoma
* History of invasive squamous cell carcinoma of the skin
* Dysplastic melanocytic nevus syndrome
* Antinuclear antibodies (ds-DNA, Ro/SSA, La/SSB)
* Autoimmune disorders such as Lupus erythematosus or Dermatomyositis
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* General poor health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Modified PASI (psoriasis area and severity index) | 12 months

SECONDARY OUTCOMES:
Patient visual analogue (VAS) score for therapeutic effect and severity of skin lesions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University, Department of Dermatology, Graz, Austria